CLINICAL TRIAL: NCT04040621
Title: A PHASE 1, OPEN-LABEL, SINGLE-DOSE STUDY TO ASSESS THE PHARMACOKINETICS, SAFETY AND TOLERABILITY OF CEFTAZIDIME-AVIBACTAM (CAZ-AVI) IN CHILDREN FROM 3 MONTHS TO LESS THAN 18 YEARS OF AGE WHO ARE HOSPITALIZED AND RECEIVING SYSTEMIC ANTIBIOTIC THERAPY FOR SUSPECTED OR CONFIRMED NOSOCOMIAL PNEUMONIA, INCLUDING VENTILATOR-ASSOCIATED PNEUMONIA
Brief Title: Single-dose PK Study of Ceftazidime-Avibactam In Hospitalized Children Receiving Systemic Antibiotics for Nosocomial Pneumonia
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Following regulatory consultation, the Sponsor has decided to terminate the study and analyze the current dataset. The decision to terminate was solely based on a business decision, not due to safety concerns.
Sponsor: Pfizer (Industry)
Collaborators: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: C3591025; 2018-002841-12 (EudraCT Number); EMBA (Other: Alias Study Number)
Record Dates: First submitted 2019-07-26; First posted 2019-08-01 (Actual); Results first posted 2022-09-09 (Actual); Last update posted 2022-09-09 (Actual); Status verified 2022-03

CONDITIONS: Hospitalized Children With Suspected or Confirmed Nosocomial Pneumonia
Keywords: nosocomial pneumonia, NP
MeSH Terms: conditions — Healthcare-Associated Pneumonia | interventions — avibactam, ceftazidime drug combination

STUDY DESIGN:
Intervention Model Description: Non-randomized, single arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ceftazidime-avibactam (Experimental): This arm includes 4 cohorts
  Interventions: Drug: Ceftazidime-avibactam

INTERVENTIONS:
Drug: Ceftazidime-avibactam — Single intravenous infusion of ceftazidime-avibactam over 2 hours. Dosage will vary depending upon age, weight and renal function.

SUMMARY:
This is a multicenter, multinational, open label single dose pharmacokinetic (PK) study enrolling at least 32 subjects. The study aims to characterize the pharmacokinetics (PK) of a single intravenous dose of CAZ AVI in pediatric subjects aged 3 months to less than 18 years who are receiving systemic antibiotic therapy for suspected or confirmed nosocomial pneumonia, including ventilator associated pneumonia.

DETAILED DESCRIPTION:
This is a multicenter, multinational, open label single dose pharmacokinetic (PK) study enrolling at least 32 subjects. The study aims to characterize the PK of CAZ AVI and assess its safety and tolerability following a single intravenous (IV) infusion. Subjects will be hospitalized pediatric patients who are receiving systemic antibiotic therapy for suspected or confirmed nosocomial pneumonia (NP), including ventilator associated pneumonia (VAP). The study will consist of a Screening visit (Visit 1, Day 1), during which consent will be obtained and subject eligibility will be confirmed, a Baseline/Treatment visit (Visit 2, Day 1) during which subjects will receive a single IV infusion of CAZ AVI, and then two follow up assessment visits at 24 hours (Visit 3, Day 2) and 48 hours (Visit 4, Day 3). Blood samples for PK analyses (0.5 mL per sample) will be obtained over 22 hours for Cohort 1 (7 samples), over 13 hours for Cohort 2 (6 samples), and over 6 hours for Cohorts 3 and 4 (4 samples). Additionally, for subjects who are undergoing bronchoalveolar lavage (BAL) for clinical purposes and for whom informed consent is obtained specifically for BAL, an epithelial lining fluid (ELF) sample will be collected for estimation of CAZ AVI concentrations.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following inclusion criteria to be eligible for enrollment into the study:

1. Evidence of a personally signed and dated informed consent document indicating that the subject's parent(s), legal guardian, or legally acceptable representative has been informed of all pertinent aspects of the study. As appropriate per local requirements informed assent of subjects must also be documented.
2. Willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.
3. Male or female children age ≥3 months to <18 years at Screening:

   1. Cohort 1: age 12 years to <18 years;
   2. Cohort 2: age 6 years to <12 years;
   3. Cohort 3: age 2 years to <6 years;
   4. Cohort 4: age 3 months to <2 years (must be born ≥37 weeks gestational age).
4. Hospitalized, receiving systemic antibiotic therapy for the treatment of a suspected or confirmed HAP or VAP meeting the following criteria, and expected to require hospitalization until after the follow up evaluations are completed on Day 3 (48 hours after the end of infusion):

   1. Onset of symptoms ≥48 hours after admission or <7 days after discharge from an inpatient acute or chronic care facility;
   2. New or worsening infiltrate on chest X ray;
   3. At least 1 of the following systemic signs prior to the initiation of treatment for Nosocomial Pneumonia:

   i. Fever (temperature >38°C) or hypothermia (rectal/core temperature <35°C); ii. White blood cell (WBC) count >10,000 cells/mm3, or WBC count <4,500 cells/mm3, or >15% band forms.

   d. At least 2 of the following respiratory signs or symptoms: i. A new onset of cough (or worsening of cough). ii. Production of purulent sputum or endotracheal secretions. iii. Auscultatory findings consistent with pneumonia/pulmonary consolidation (eg, rales, rhonchi, bronchial breath sounds, dullness to percussion, egophony).

   iv. Dyspnea, tachypnea or hypoxemia (O2 saturation <90% or PaO2 <60 mmHg while breathing room air).

   v. A need for mechanical ventilation or, for already ventilated subjects, acute changes made in the ventilator support system to enhance oxygenation, as determined by, for example arterial blood gas or worsening PaO2/FiO2.
5. Likely to survive the current illness or hospitalization.
6. Sufficient IV access (peripheral or central) to receive study drug and dedicated access for PK sampling.

Exclusion Criteria:

Subjects with any of the following characteristics/conditions will not be included in the study:

1. Investigator site staff members directly involved in the conduct of the study and their family members, site staff members otherwise supervised by the Investigator, or subjects who are Pfizer employees, including their family members, directly involved in the conduct of the study.
2. Participation in other studies involving investigational drug(s) within 30 days prior to study entry and/or during study participation.
3. Other acute or chronic medical or psychiatric condition including recent (within the past year) or active suicidal ideation or behavior or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the Investigator, would make the subject inappropriate for entry into this study.
4. Past or current history of epilepsy or seizure disorder (excluding childhood febrile seizures.
5. Severe renal impairment defined as creatinine clearance (CrCL) ≤30 mL/min/1.73 m2 calculated using the child's measured height (length) and serum creatinine with the Bedside Schwartz equation (Schwartz, Munoz, et al., 2009):3 CrCL (mL/min/1.73 m2) =
6. Documented history of any hypersensitivity or allergic reaction to any β lactam antibiotic.
7. Pregnant female subjects; breastfeeding female subjects; fertile male subjects and female subjects of childbearing potential who are unwilling or unable to use a highly effective method of contraception as outlined in this protocol for the duration of the study and for at least 28 days after the last dose of CAZ AVI.
8. Acute hepatitis in the prior 6 months, a prior history of cirrhosis, acute hepatic failure, or acute decompensation of chronic hepatic failure; and/or any of the following blood test results, for any individual, when assessed for eligibility:

   1. Bilirubin >3 × upper limit of normal (ULN), unless isolated hyperbilirubinemia is directly related to the acute infection or due to known Gilbert's disease;
   2. ALT or AST >3 × ULN values used by the laboratory performing the test. Subjects with values >3 × ULN and <5 × ULN are eligible if this value is acute and directly related to the infectious process being treated. This must be documented;
   3. ALP >3 × ULN. Subjects with values >3 × ULN and <5 × ULN are eligible if this value is acute and directly related to the infectious process being treated. This must be documented.
9. Any condition (eg, septic shock, burns, cystic fibrosis, acute hemodynamic instability, including those conditions not responding to pressor support) that would make the patient, in the opinion of the Investigator, unsuitable for the study (eg, would place a patient at risk; compromise the quality of the data; or interfere with the absorption, distribution, metabolism, or excretion of CAZ AVI).
10. Receipt of a blood or blood component or scheduled for transfusion within the PK sampling period (eg, red blood cells, fresh frozen plasma, platelets) transfusion during the 24 hour period before enrollment.
11. Body mass index (BMI) below the 5th percentile or above the 95th percentile for height, age, and weight except for children <2 years of age as BMI is not considered a screening tool for healthy weight in children under 2 years of age.
12. Treatment with ceftazidime within 12 hours of CAZ AVI administration or treatment with ceftazidime within 24 hours of CAZ AVI administration in subjects with renal impairment (CrCL ≤50 mL/min/1.73 m2).
13. Treatment with potent inhibitors of OAT1 and/or OAT3 (eg, probenecid, p aminohippuric acid (PAH), or teriflunomide).

Ages: 3 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 4 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2021-04-09 (Actual); Study Completion 2021-05-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (4):
- China (2):
  - Wuxi Children's Hospital, Wuxi, Jiangsu
  - Chengdu Women's and Children's Central Hospital, Chengdu, Sichuan
- Taiwan (2):
  - Taipei Municipal Wanfang Hospital, Taipei
  - Chang Gung Memorial Hospital-Linkou, Taoyuan

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C3591025

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Hospitalized pediatric participants who were receiving systemic antibiotic therapy for suspected or confirmed nosocomial pneumonia (NP), including ventilator-associated pneumonia (VAP) were enrolled.
Pre-assignment Details: Only 4 participants were enrolled before trial was stopped prematurely. Data was planned to be reported per cohort but doing so would risk re-identification of participants. Only participant flow and baseline characteristics data are reported for all enrolled participants as 1 reporting group.
Groups:
- All Enrolled Participants: Ceftazidime-Avibactam (CAZ-AVI): Participants received 50 milligram (mg) per kilogram (kg) of CAZ and 12.5 mg/kg of AVI intravenously on Day 1.
Period: Overall Study
Arm/Group | All Enrolled Participants: Ceftazidime-Avibactam (CAZ-AVI)
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The safety analysis set included all participants who received any amount of IV study dose of CAZ AVI.
Groups:
- All Enrolled Participants: Ceftazidime-Avibactam (CAZ-AVI): Participants received 50 mg/kg of CAZ and 12.5 mg/kg of AVI intravenously on Day 1.
Arm/Group | All Enrolled Participants: Ceftazidime-Avibactam (CAZ-AVI)
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Plasma Concentration Time Summary for Ceftazidime and Avibactam
Time Frame: Day 1: 2, 2.25, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 13, 24 hours post dose
Population: Pharmacokinetics (PK) analysis set included all participants who received a complete IV study dose of CAZ-AVI and had at least 1 ceftazidime and/or avibactam plasma measurement available. Planned analysis was to report data cohort wise. Due to low enrolment providing data per cohort would risk re-identification of participants. Hence, data are not reported.
Arm/Group | All Enrolled Participants: Ceftazidime-Avibactam (CAZ-AVI)
Number analyzed (Participants) | 0

2. Primary Outcome: Area Under the Plasma Concentration-Time Profile From Time 0 to 8 Hours (AUC0-8 Hours)
Time Frame: Day 1: 2, 2.25, 2.5, 3, 3.5, 4, 5, 6, 8 hours post dose
Population: PK analysis set included all participants who received a complete IV study dose of CAZ-AVI and had at least 1 ceftazidime and/or avibactam plasma measurement available. Planned analysis was to report data cohort wise. Due to low enrolment providing data per cohort would risk re-identification of participants. Hence, data are not reported.
Arm/Group | All Enrolled Participants: Ceftazidime-Avibactam (CAZ-AVI)
Number analyzed (Participants) | 0

3. Primary Outcome: Area Under the Curve From Time Zero to Extrapolated Infinite Time of CAZ-AVI (AUCinf)
Description: AUCinf = AUClast + (Clast*/ kel), where Clast* is the estimated concentration at the time of the last quantifiable concentration and kel is the terminal phase rate constant calculated by a linear regression of the log-linear concentration-time curve.
Time Frame: Day 1: 2, 2.25, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 13, 24 hours post dose
Population: as for outcome 2
Arm/Group | All Enrolled Participants: Ceftazidime-Avibactam (CAZ-AVI)
Number analyzed (Participants) | 0

4. Primary Outcome: Area Under the Concentration-Time Profile From Time 0 to Time to Last Quantifiable Concentration (AUClast) of CAZ-AVI
Time Frame: Day 1: 2, 2.25, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 13, 24 hours post dose
Population: as for outcome 2
Arm/Group | All Enrolled Participants: Ceftazidime-Avibactam (CAZ-AVI)
Number analyzed (Participants) | 0

5. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of CAZ-AVI
Time Frame: Day 1: 2, 2.25, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 13, 24 hours post dose
Population: as for outcome 2
Arm/Group | All Enrolled Participants: Ceftazidime-Avibactam (CAZ-AVI)
Number analyzed (Participants) | 0

6. Primary Outcome: Time to Last Quantifiable Plasma Concentration (Tlast) of CAZ-AVI
Time Frame: Day 1: 2, 2.25, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 13, 24 hours post dose
Population: as for outcome 2
Arm/Group | All Enrolled Participants: Ceftazidime-Avibactam (CAZ-AVI)
Number analyzed (Participants) | 0

7. Primary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of CAZ-AVI
Time Frame: Day 1: 2, 2.25, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 13, 24 hours post dose
Population: as for outcome 2
Arm/Group | All Enrolled Participants: Ceftazidime-Avibactam (CAZ-AVI)
Number analyzed (Participants) | 0

8. Primary Outcome: Termination Elimination Half-Life (t1/2) of CAZ-AVI
Time Frame: Day 1: 2, 2.25, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 13, 24 hours post dose
Population: as for outcome 2
Arm/Group | All Enrolled Participants: Ceftazidime-Avibactam (CAZ-AVI)
Number analyzed (Participants) | 0

9. Primary Outcome: Clearance (CL) of CAZ-AVI
Description: Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood (rate at which a drug is metabolized or eliminated by normal biological processes). Clearance obtained after intravenous infusion dose (apparent clearance) is influenced by the fraction of the dose absorbed. CL = Dose/AUCinf.
Time Frame: Day 1: 2, 2.25, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 13, 24 hours post dose
Population: as for outcome 2
Arm/Group | All Enrolled Participants: Ceftazidime-Avibactam (CAZ-AVI)
Number analyzed (Participants) | 0

10. Primary Outcome: Volume of Distribution of CAZ-AVI
Description: Volume of distribution at steady state (Vss) = Clearance (CL) × Mean Residence Time (MRT), MRT = Area under the first moment curve from 0 time to infinity (AUMCinf)/AUCinf - (infusion time/2), AUMCinf = AUMClast + (t × Cest1*/kel) +(Cest1*/kel2), 1Cest = e(-KEL × Tlast) × KELC0 , where C0 is the back-extrapolated concentration at time zero.
Time Frame: Day 1: 2, 2.25, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 13, 24 hours post dose
Population: as for outcome 2
Arm/Group | All Enrolled Participants: Ceftazidime-Avibactam (CAZ-AVI)
Number analyzed (Participants) | 0

11. Primary Outcome: Volume of Distribution During Terminal Phase (Vz) of CAZ-AVI
Description: Vz = Dose/(AUCinf × kel).
Time Frame: Day 1: 2, 2.25, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 13, 24 hours post dose
Population: as for outcome 2
Arm/Group | All Enrolled Participants: Ceftazidime-Avibactam (CAZ-AVI)
Number analyzed (Participants) | 0

12. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Time Frame: Day 1 up to maximum of 35 days after last dose of study treatment (maximum of 36 days)
Population: Safety set included all participants who had received any amount of IV study dose of CAZ AVI. Planned analysis was to report data cohort wise. Due to low enrolment providing data per cohort would risk re-identification of participants. Hence, data are not reported.
Arm/Group | All Enrolled Participants: Ceftazidime-Avibactam (CAZ-AVI)
Number analyzed (Participants) | 0

13. Secondary Outcome: Number of Participants With Death and Discontinuations Due to Adverse Events (AEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship.
Time Frame: Day 1 up to maximum of 35 days after last dose of study treatment (maximum of 36 days)
Population: as for outcome 12
Arm/Group | All Enrolled Participants: Ceftazidime-Avibactam (CAZ-AVI)
Number analyzed (Participants) | 0

14. Secondary Outcome: Number of Participants With Clinically Significant Abnormal Laboratory Values
Description: Following parameters were analyzed for laboratory examination: Clinical Chemistry-sodium, potassium, chloride, bicarbonate, creatinine, blood urea nitrogen, glucose-non fasting, calcium, phosphorus, magnesium, alkaline phosphatase, gamma glutamyl transferase, aspartate transaminase, alanine transaminase, creatinine kinase, lactate dehydrogenase, indirect bilirubin, total bilirubin; Hematology- hematocrit, hemoglobin, red blood cells (RBC), white blood cells (WBC), neutrophils, lymphocytes, monocytes, eosinophils, basophils, neutrophils immature, platelets, mean cell volume, mean cell hemoglobin, β- human chorionic gonadotropin (hCG) pregnancy test (blood or urine) for females; Urinalysis- appearance (color, clarity), bilirubin, glucose, ketones leukocyte esterase, nitrite, pH, protein, specific gravity, urobilinogen, microscopic (RBC, WBC, casts, crystals, bacteria, yeast, parasites).
Time Frame: Baseline up to Day 3
Population: as for outcome 12
Arm/Group | All Enrolled Participants: Ceftazidime-Avibactam (CAZ-AVI)
Number analyzed (Participants) | 0

15. Secondary Outcome: Number of Participants With Clinically Significant Physical Examination Abnormalities
Description: Parameters assessed for physical examination included: body weight and height. Abnormality was judged by investigator.
Time Frame: Baseline up to Day 3
Population: Safety set included all participants who had received any amount of IV study dose of CAZ-AVI.Planned analysis was to report data cohort wise. Due to low enrolment providing data per cohort would risk re-identification of participants. Hence, data are not reported.
Arm/Group | All Enrolled Participants: Ceftazidime-Avibactam (CAZ-AVI)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Day 1 up to maximum of 35 days after last dose of study treatment (maximum of 36 days)
Description: Data cannot be reported because doing so would risk re-identification of participants.
Arm/Group | All Enrolled Participants: Ceftazidime-Avibactam (CAZ-AVI)
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 0/4

LIMITATIONS AND CAVEATS:
Only 4 participants were enrolled in this study. Outcome measures and AE data were not reported by cohort as planned in the protocol because doing so would risk re-dentification of the individual participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2019-06-12): https://cdn.clinicaltrials.gov/large-docs/21/NCT04040621/Prot_000.pdf
  • Statistical Analysis Plan (2019-08-02): https://cdn.clinicaltrials.gov/large-docs/21/NCT04040621/SAP_001.pdf